CLINICAL TRIAL: NCT05930613
Title: Efficacy of Certolizumab in Women With Unexplained Recurrent Implantation Failure: a Double-blind Randomized Controlled Trial
Brief Title: Certolizumab in Recurrent Implantation Failure (RIF)
Acronym: CERTIFY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200031; 2021-005309-28 (EudraCT Number)
Record Dates: First submitted 2023-05-22; First posted 2023-07-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Unexplained Implantation Failure
Keywords: Recurrent Implantation Failure; Immunomodulation; Anti-TNF-α; Certolizumab; Pregnancy
MeSH Terms: interventions — Certolizumab Pegol; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Certolizumab (CIMZIA® ; TNF-α antagonist )
  Interventions: Drug: Certolizumab (CIMZIA® ; TNF-α antagonist)
- 2 (Placebo Comparator): Placebo (NaCl 0.9 % solution)
  Interventions: Drug: Placebo (NaCl 0.9 % solution)

INTERVENTIONS:
Drug: Certolizumab (CIMZIA® ; TNF-α antagonist) — 400mg of certolizumab injected subcutaneously monthly from 5 weeks before embryo transfer until 7 weeks of gestation (injections at 5 and 1 week before embryo transfer, 3 and 7 weeks after embryo transfer) for a total of 4 injections in case of ongoing intrauterine pregnancy.
  Arms: 1
Drug: Placebo (NaCl 0.9 % solution) — NaCl 0,9% injected subcutaneously monthly from 5 weeks before embryo transfer until 7 weeks of gestation (injections at 5 and 1 week before embryo transfer, 3 and 7 weeks after embryo transfer) for a total of 4 injections in case of ongoing intrauterine pregnancy.
  Arms: 2

SUMMARY:
Recurrent implantation failure (RIF), defined as the absence of clinical pregnancy after the transfer of three good-quality embryos, concerns up to 40% of IVF couples and is associated with a low success rate. The causes remain unexplained in over 50% of cases.

Various dysimmune changes (related to immune T cells profiles, pro-inflammatory cytokines levels) have been described in unexplained RIF as compared to fertile controls, and it has been estimated that such dysimmunity may occur in 50% of unexplained RIFs. Previous data on a benefit of general immune modulation by steroids or immunoglobulins are heterogenous and failed to demonstrate clinically significant benefit. The proinflammatory cytokine Tumor Necrosis Factor (TNF) α participates in the regulation of the immune balance of the endometrium, its peripheral blood and endometrial concentrations are increased in RIF patients as compared to fertile controls. In 2009, a pilot placebo controlled study showed that TNF-α antagonist treatment allowed a 56% live birth rate (versus 13% in controls) in 13 women with unexplained RIF. Due to the lack of maternal and fetal tolerance data, TNF-α antagonists were not further evaluated. Today, safety data issued from 1200 pregnancies are reassuring allowing the use of TNF-α antagonists during pregnancy (www.lecrat.org). In addition the TNF-α antagonist certolizumab does not cross the placental barrier.

We hypothesize that certolizumab may improve clinical pregnancy rates in women with unexplained RIF with a good safety profile.

DETAILED DESCRIPTION:
The European Society of Human Reproduction and Embryology (ESHRE) consortium has proposed to define recurrent implantation failure (RIF) as the failure to obtain a clinical pregnancy after the transfer of three good-quality embryos according to the Istanbul consensus 2011. Although its prevalence is difficult to estimate, RIF could concern up to 40% of couples undergoing assisted reproductive technology (ART) treatments. More than 50% of RIF cases remain unexplained after extensive exploration and clinical pregnancy rate in this population is particularly low, estimated at about 15%.

Endometrial environment plays a crucial role in embryo implantation and early placental development. In normal pregnancy, the survival of the semi-allogeneic fetus is dependent on the induction of maternal immune tolerance, with regulatory T cells and Th-2 anti-inflammatory profile. Several studies show a misbalance of immune cells and cytokines expression in women with implantation failure. Most studies analyze immune cells and cytokines profile in peripheral blood, with few data on cells and cytokines profiles in endometrial tissues during the periimplantation period. However, the immune endometrial balance could be disturbed in up to 80% of RIF cases.

Tumor Necrosis Factor (TNF) α, together with other pro-inflammatory cytokines, participates in the regulation of the immune balance of the endometrium. TNF-α and TNF-α / interleukin (IL)-10 ratio are increased in the endometrium of RIF patients, which suggests they could be involved in physiopathology of RIF.

To date there is no effective treatment to improve the low clinical pregnancy rate in unexplained RIF. The repeated failure of embryo transfers and the lack of efficient treatment are associated with psychological distress in infertile couples and raises economic problems because of the important cost of in vitro fertilisation (IVF).

Some treatments with immunomodulatory effect, such as steroids, were previously evaluated. However, studies were small and included heterogeneous populations, resulting in inconclusive results.

Our hypothesis is that TNF-α antagonists may be particularly useful by blocking TNF-α induced excessive immune-response.

In a pilot placebo controlled study, TNF-α antagonists were associated with 56% live births versus 13% in controls, in 13 women with unexplained implantation failure. However, this treatment was not further evaluated in this indication because of the lack of tolerance data and the fear of congenital abnormalities.

Concerning the safety of TNF-α antagonists, we now have sufficient data as they are widely used since more than 15 years in several autoimmune and inflammatory diseases. More than 1200 women treated with TNF-α antagonists for an inflammatory disease have provided evidence of their safety in early pregnancy and the French national center of drug-related effects (www.lecrat.org) allows the use of TNF-α antagonists during pregnancy, except during the third trimester. Among TNF-α antagonists, certolizumab have the particularity not to cross the placental barrier and thus can be used during pregnancy, This is why we focus on this particular drug for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Idiopathic, male or tubal factor infertility
* Unexplained recurrent implantation failure defined as consecutive failure to obtain clinical pregnancy after at least transfers of 3 good-quality embryos (Istanbul criteria)
* Affiliation to a French social security system (beneficiary or legal)
* Informed and signed consent

Exclusion Criteria:

Known cause of RIF among the following:

* Genetic parental anomalies
* Non-gestational diabetes mellitus of type I and II,
* Infectious disease
* Antiphospholipid syndrome
* Sickle cell disease
* Diffuse adenomyosis
* No contraindication to Freeze-thaw embryo transfer (FET) treatment

Linked to certolizumab:

* Hypersensitivity to the active substances or to any of the excipients
* Primary or secondary immunodeficiency (history of or currently active)
* Active uncontrolled infection
* Active tuberculosis
* Cardiac insufficiency (moderate to severe, New York Heart Association (NYHA) III/IV classes)
* Any malignant neoplasm except adequately treated basal or squamous cell carcinoma of the skin
* Immunization with a live/ attenuated vaccine within 4 weeks prior to baseline or simultaneously with treatment
* Cytopenia as defined by platelet count < 100 × 109/L (100,000/mm3), hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L), absolute neutrophil count < 2.0 × 109/L (2000/mm3), lymphocyte count < 0.5 × 109/L (500/mm3)
* Liver cytolysis (AST / ALT > 5 N)
* Insufficient kidney function, as defined by a serum creatinine of more than 3 mg/dL or creatinine clearance of 20 ml/min or less
* Demyelinating neurological disease

Linked to rifampicin and isoniazid (RIFINAH®)

* Hypersensitivity to the active substances or to any of the excipients
* Porphyria
* Decreased blood-clotting from low vitamin K
* Liver cytolysis (AST / ALT >5 N)
* Combination with bictegravir, cobicistat, daclatasvir, dasabuvir, delamanid, grazoprevir / elbasvir, protease inhibitors boosted by ritonavir, isavuconazole, ledipasvir, lurasidone, midostaurine, ombitasvir / paritaprévir, praziquantel, rilpivirine, sofosbuvir, velpatasvir, voriconazole, voxilaprevir
* Acute hepatitis, hepatic failure or chronic hepatic disease
* Acute nephropathy

Contraindication to anti-pneumococcal vaccination (Pneumovax®)

- Hypersensitivity to the active substances or to any of the excipients

Other criteria:

* Absence of health insurance (include AME)
* Subject under guardianship or curatorship
* Subject deprived of their liberty by a judicial or administrative decision
* Participation in another interventional study or being in the exclusion period at the end of a previous study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy defined as the presence of cardiac activity on ultrasound scan | 5 weeks +/- 6 days of gestation
  Presence of cardiac activity on ultrasound scan at 5 weeks +/- 6 days of gestation

SECONDARY OUTCOMES:
Live birth | 22 to 40 weeks of gestation
Miscarriage | Before 12 weeks of gestation
  Miscarriage defined as spontaneous abortion or pregnancy stop
All adverse events distinguishing serious adverse events | Through study completion, a maximum of 64 months and 3 weeks
  Adverse events of interest are :
  * multiple pregnancies
  * ectopic pregnancy
  * fetal abnormalities
  * small for gestational age
  * intrauterine growth restriction
  * preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Arsene MEKINIAN, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint-Antoine Hospital - APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.